CLINICAL TRIAL: NCT04135144
Title: Comparison of the Effects of Two Different Home Exercise Programs in Neck Pain
Brief Title: Different Home Exercise Programs in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Özden Laçin (Other)
Responsible Party: Sponsor-Investigator, Özden Laçin, Principal Investigator, Istanbul Arel University
Organization: Istanbul Arel University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ozdenyasarer
Record Dates: First submitted 2019-10-14; First posted 2019-10-22 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Neck Pain; Exercise Training
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (printed materials), (Active Comparator): Group 1 was given home exercise method with printed materials
  Interventions: Other: Group 1 (printed materials)
- Group 2 (video phone reminder) (Active Comparator): Group 2 was given exercise with home exercise method with video phone reminder
  Interventions: Other: Group 2 (video phone reminder)

INTERVENTIONS:
Other: Group 1 (printed materials) — Exercises were given at least 3 times a week for 10 weeks and 1 set per day for a total of 6 weeks. individuals; normal joint movement exercises; neck flexion, lateral flexion, rotation, extension and retraction movements, isometric exercises; neck flexion, extension, lateral flexion and rotation movements and stretching exercises; neck lateral flexion, neck rotation and flexion movements were given.
  Other Names: home exercise with printed materials
  Arms: Group 1 (printed materials),
Other: Group 2 (video phone reminder) — Exercises were given at least 3 times a week for 10 weeks and 1 set per day for a total of 6 weeks. individuals; normal joint movement exercises; neck flexion, lateral flexion, rotation, extension and retraction movements, isometric exercises; neck flexion, extension, lateral flexion and rotation movements and stretching exercises; neck lateral flexion, neck rotation and flexion movements were given.
  Other Names: home exercise with video phone reminder
  Arms: Group 2 (video phone reminder)

SUMMARY:
Purpose: The aim of this study was to compare the effects of two different home exercise methods on exercise compliance, neck pain and neck disability in individuals with neck pain.

Material and metods: The study, carried out between February 2018 and May 2018 at Istanbul Arel University Vocational School, was performed with 60 people aged 25-60 years who were suffering from neck pain in academic and administrative staff. The cases were randomly divided into two groups. In Group 1, the case was given home exercise method (B.M.E.Y) with printed materials whereas Group 2 was given exercise with home exercise method (V.H.E.Y) with video phone reminder. Pain intensity was evaluated before and after exercise with 'Visual Analog Scale' (VAS), whereas the level of neck disability was evaluated before and after exercise with 'Neck Pain and Disability Score' (NPDS). The obtained results were analyzed using appropriate statistical methods.

DETAILED DESCRIPTION:
Both groups were prescribed the same type of exercise, duration of exercise and number of repetitions. group 1 completed the exercise program and marked the exercise attendance schedule. At the end of the program, these charts were collected from the subjects and the continuity was evaluated. The group marked the exercises completed with 2 phone app. In the program used, exercise continuity of the cases was evaluated as days.

Exercises were given at least 3 times a week for 10 weeks and 1 set per day for a total of 6 weeks. individuals; normal joint movement exercises; neck flexion, lateral flexion, rotation, extension and retraction movements, isometric exercises; neck flexion, extension, lateral flexion and rotation movements and stretching exercises; neck lateral flexion, neck rotation and flexion movements were given.

ELIGIBILITY:
Inclusion Criteria:

* complaint of neck pain,
* Being between 25-60 years of age

Exclusion Criteria:

* taking painkillers regularly,
* undergoing any neck surgery and severe trauma,
* presence of any diagnosed neck disease

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Neck disability | 6 weeks
  Self reported. The level of neck disability was evaluated before and after exercise with 'Neck Pain and Disability Score' . Each question is measured on a scale from 0 (no disability) to 5, and an overall score out of 100 is calculated by adding each item score together.
Pain intensity | 6 weeks
  Self reported pain intensity .. Pain intensity was evaluated before and after exercise with 'Visual Analog Scale'. Each item scored is 0-10 (0=no pain 10=pain as bad as can be)

CONTACTS AND LOCATIONS:
Overall Officials: Özden Laçin, Study Director — İstanbul Arel Uiversity
Locations (1):
- İstanbul Arel University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Yasarer O, Yilmaz HG, Dogan H. Comparison of two different delivery methods of home-based exercise on neck pain. Somatosens Mot Res. 2024 Dec;41(4):205-212. doi: 10.1080/08990220.2023.2194389. Epub 2023 Apr 7. PMID 37026597